CLINICAL TRIAL: NCT02389959
Title: Intranasal Bevacizumab for HHT-Related Epistaxis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Peter Hwang, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 29501
Record Dates: First submitted 2015-03-11; First posted 2015-03-17 (Estimated); Results first posted 2021-02-15 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: HHT; Hereditary Hemorrhagic Telangiectasia; Epistaxis; Nose Bleeds; Nasal Bleeding
Keywords: HHT; Hereditary Hemorrhagic Telangiectasia; epistaxis; nose bleeds; nasal bleeding; Avastin; bevacizumab
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Epistaxis | interventions — Bevacizumab; Sodium Chloride; Fluoridation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bevacizumab (Experimental): The Stanford Hospital Investigational Pharmacy will perform all randomization, drug storage and management, as well as mixing and packaging for double-blinded injection of bevacizumab or saline control. Patients will undergo standard-of-care bipolar electrocautery of nasal telangiectasias in the Stanford Surgery Center operating room. At the time of electrocautery, patients will receive intranasal injection of either study drug or saline control. The surgeon performing the injection will be blinded to whether injection is composed of bevacizumab or saline control. Bevacizumab will be mixed by the Stanford Hospital Pharmacy to a total dose of 100mg in 4mL, and 50mg (2mL) will be injected into each side of the nose. Injections will be performed according to the standardized four-point injection protocol (0.5mL/site) based on the vascular anatomy of the nose published in 2012 by Dheyauldeen et al.
  Interventions: Drug: Bevacizumab
- Saline Control (Placebo Comparator): The Stanford Hospital Investigational Pharmacy will perform all randomization, drug storage and management, as well as mixing and packaging for double-blinded injection of bevacizumab or saline control. Patients will undergo standard-of-care bipolar electrocautery of nasal telangiectasias in the Stanford Surgery Center operating room. At the time of electrocautery, patients will receive intranasal injection of either study drug or saline control. The surgeon performing the injection will be blinded to whether injection is composed of bevacizumab or saline control. The saline control placebo will be mixed by the Stanford Hospital Pharmacy to a total dose of 4mL in order to be identical in quantity and appearance to the mixed doses of bevacizumab, and 2mL will be injected into each side of the nose. Injections will be performed according to the standardized four-point injection protocol (0.5mL/site) based on the vascular anatomy of the nose published in 2012 by Dheyauldeen et al.
  Interventions: Drug: Placebo (Saline)

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab will be mixed by the Stanford Hospital Pharmacy to a total dose of 100mg in 4mL, and 50mg (2mL) will be injected into each side of the nose
  Other Names: Avastin
  Arms: Bevacizumab
Drug: Placebo (Saline) — 4mL of saline will be mixed by the Stanford Hospital Pharmacy as a control
  Other Names: Salt water
  Arms: Saline Control

SUMMARY:
This is a randomized, controlled, double-blind, placebo-controlled trial of intranasal Avastin (bevacizumab) injection versus saline control for control of HHT-related epistaxis when used in conjunction with bipolar electrocautery.

DETAILED DESCRIPTION:
Hereditary hemorrhagic telangiectasia (HHT) is an autosomal dominant genetic disorder characterized by systemic vascular malformations that result from mutations of the ENG gene, which encodes for factors in the vascular endothelial growth factor (VEGF) pathway. HHT is diagnosed by the Curacao Criteria including the presence of epistaxis; telangiectasias or vascular malformations in the lungs, liver, or nervous system; and a positive family history involving a first-degree relative. One of the most common presentations of this disease is recurrent and profound epistaxis, with many patients reporting more than 4 epistaxis episodes in a day, many lasting up to an hour. HHT-related epistaxis often results in severe anemia requiring intravenous iron and repeated blood transfusions, and also carries significant psychosocial disability relating to impaired quality of life and work absenteeism. Multiple approaches to treatment have been described, including electrocautery, laser treatment, embolization, septodermoplasty, and as a last resort, Young's procedure, involving closure of the nasal vestibule. These approaches are largely palliative, with variable effectiveness, and almost always require repeated procedures for chronic management of bleeding. There is a great need for the development of new treatment options for reducing the medical morbidity and quality of life impairment associated with refractory epistaxis in HHT.

Recently there has been promising data suggesting that inhibition of angiogenesis may be an effective strategy for managing HHT-related bleeding. Circulating concentrations of VEGF are significantly elevated in HHT, making VEGF an attractive therapeutic target. Preliminary studies suggest that bevacizumab, a recombinant monoclonal antibody that inhibits the biologic activity of VEGF, can significantly improve epistaxis severity when topically applied, locally injected, or intravenously administered. However, these early pilot studies of bevacizumab have been limited exclusively to retrospective case series. As yet, there has been no prospective double-blind placebo controlled trial with serial follow up time points to establish the role of bevacizumab in the treatment of HHT-related epistaxis.

Based on existing level 4 evidence that suggests that bevacizumab injection is beneficial in the management of HHT-related epistaxis, we hypothesize that patients who receive intranasal injection with bevacizumab at the time of electrocautery treatment will have an improvement in the frequency and severity of epistaxis compared to patients who receive injection of saline control.

ELIGIBILITY:
Inclusion Criteria:

1. The patient carries a diagnosis of hereditary hemorrhagic telangiectasia (HHT)
2. The patient is to undergo treatment with electrocautery in the operating room under endoscopic visualization
3. The patient is able to give informed consent
4. The patient is at least 18 years old

Exclusion Criteria:

1. The patient has had prior treatment with systemic or nasal bevacizumab within the past year
2. The patient has undergone electrocautery for epistaxis within the 6 months prior to study enrollment
3. The patient is a minor
4. The patient is pregnant
5. The patient is incapable of understanding the consent process
6. The patient has a history of HIV or another known cause of immunosuppression, or is actively taking immunosuppressive medications due to organ transplantation, rheumatoid disease, or other medical conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-08-04 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter H Hwang, MD, Principal Investigator — Stanford University, Department of Otolaryngology- Head and Neck Surgery
Locations (1):
- Stanford University Department of Otolaryngology- Head and Neck Surgery, Stanford, California, United States

REFERENCES:
- [Background] Shovlin CL, Guttmacher AE, Buscarini E, Faughnan ME, Hyland RH, Westermann CJ, Kjeldsen AD, Plauchu H. Diagnostic criteria for hereditary hemorrhagic telangiectasia (Rendu-Osler-Weber syndrome). Am J Med Genet. 2000 Mar 6;91(1):66-7. doi: 10.1002/(sici)1096-8628(20000306)91:13.0.co;2-p. PMID 10751092
- [Background] Lund VJ, Howard DJ. A treatment algorithm for the management of epistaxis in hereditary hemorrhagic telangiectasia. Am J Rhinol. 1999 Jul-Aug;13(4):319-22. doi: 10.2500/105065899782102890. PMID 10485021
- [Background] Sadick H, Riedel F, Naim R, Goessler U, Hormann K, Hafner M, Lux A. Patients with hereditary hemorrhagic telangiectasia have increased plasma levels of vascular endothelial growth factor and transforming growth factor-beta1 as well as high ALK1 tissue expression. Haematologica. 2005 Jun;90(6):818-28. PMID 15951295
- [Background] Simonds J, Miller F, Mandel J, Davidson TM. The effect of bevacizumab (Avastin) treatment on epistaxis in hereditary hemorrhagic telangiectasia. Laryngoscope. 2009 May;119(5):988-92. doi: 10.1002/lary.20159. PMID 19194865
- [Background] Karnezis TT, Davidson TM. Efficacy of intranasal Bevacizumab (Avastin) treatment in patients with hereditary hemorrhagic telangiectasia-associated epistaxis. Laryngoscope. 2011 Mar;121(3):636-8. doi: 10.1002/lary.21415. Epub 2010 Dec 16. PMID 21344445
- [Background] Rohrmeier C, Sachs HG, Kuehnel TS. A retrospective analysis of low dose, intranasal injected bevacizumab (Avastin) in hereditary haemorrhagic telangiectasia. Eur Arch Otorhinolaryngol. 2012 Feb;269(2):531-6. doi: 10.1007/s00405-011-1721-9. Epub 2011 Jul 31. PMID 21805356
- [Background] Chen S 4th, Karnezis T, Davidson TM. Safety of intranasal Bevacizumab (Avastin) treatment in patients with hereditary hemorrhagic telangiectasia-associated epistaxis. Laryngoscope. 2011 Mar;121(3):644-6. doi: 10.1002/lary.21345. Epub 2010 Nov 11. PMID 21344447
- [Background] Dheyauldeen S, Ostertun Geirdal A, Osnes T, Vartdal LS, Dollner R. Bevacizumab in hereditary hemorrhagic telangiectasia-associated epistaxis: effectiveness of an injection protocol based on the vascular anatomy of the nose. Laryngoscope. 2012 Jun;122(6):1210-4. doi: 10.1002/lary.23303. Epub 2012 May 7. PMID 22565282
- [Background] Karnezis TT, Davidson TM. Treatment of hereditary hemorrhagic telangiectasia with submucosal and topical bevacizumab therapy. Laryngoscope. 2012 Mar;122(3):495-7. doi: 10.1002/lary.22501. Epub 2011 Dec 6. PMID 22147664
- [Background] Hoag JB, Terry P, Mitchell S, Reh D, Merlo CA. An epistaxis severity score for hereditary hemorrhagic telangiectasia. Laryngoscope. 2010 Apr;120(4):838-43. doi: 10.1002/lary.20818. PMID 20087969
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Lennox PA, Hitchings AE, Lund VJ, Howard DJ. The SF-36 health status questionnaire in assessing patients with epistaxis secondary to hereditary hemorrhagic telangiectasia. Am J Rhinol. 2005 Jan-Feb;19(1):71-4. PMID 15794078
- [Background] Ingrand I, Ingrand P, Gilbert-Dussardier B, Defossez G, Jouhet V, Migeot V, Dufour X, Klossek JM. Altered quality of life in Rendu-Osler-Weber disease related to recurrent epistaxis. Rhinology. 2011 Jun;49(2):155-62. doi: 10.4193/Rhino09.138. PMID 21743869
- [Background] Steinbrook R. The price of sight--ranibizumab, bevacizumab, and the treatment of macular degeneration. N Engl J Med. 2006 Oct 5;355(14):1409-12. doi: 10.1056/NEJMp068185. No abstract available. PMID 17021315
- [Background] Smith KA, Rudmik L. Cost collection and analysis for health economic evaluation. Otolaryngol Head Neck Surg. 2013 Aug;149(2):192-9. doi: 10.1177/0194599813487850. Epub 2013 May 2. PMID 23641023
- [Background] Koopmanschap MA. PRODISQ: a modular questionnaire on productivity and disease for economic evaluation studies. Expert Rev Pharmacoecon Outcomes Res. 2005 Feb;5(1):23-8. doi: 10.1586/14737167.5.1.23. PMID 19807557
- [Background] Brazier J, Roberts J, Deverill M. The estimation of a preference-based measure of health from the SF-36. J Health Econ. 2002 Mar;21(2):271-92. doi: 10.1016/s0167-6296(01)00130-8. PMID 11939242
- [Background] Brazier JE, Roberts J. The estimation of a preference-based measure of health from the SF-12. Med Care. 2004 Sep;42(9):851-9. doi: 10.1097/01.mlr.0000135827.18610.0d. PMID 15319610

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab: Bevacizumab mixed by the Stanford Hospital Pharmacy to a total dose of 100mg in 4mL, and 50mg (2mL), injected into each side of the nose
- Saline Control: Placebo (4mL of saline) mixed by the Stanford Hospital Pharmacy as a control.
Period: Overall Study
Arm/Group | Bevacizumab | Saline Control
Started | 20 | 20
Completed | 18 | 19
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Population: 1 participant did not complete the baseline questionnaires.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bevacizumab | Saline Control | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.37 (15.4) | 55.35 (11.75) | 52.44 (13.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 11 | 10 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 1
  Caucasian | 15 | 18 | 33
  Hispanic | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 20 | 39
Epistaxis Severity Score (ESS) [Median (Inter-Quartile Range); unit: units on a scale] — ESS is a standardized and reproducible outcome measure for the control of epistaxis. It is composed of six factors that are independent predictors of self-described epistaxis severity. The range is 0 to 13. The higher the score worse is epistaxis severity.
  units on a scale | 5.83 [3.91 to 6.79] | 5.06 [3.21 to 7.01] | 5.35 [3.51 to 6.90]
SF-12 Physical Component Summary (PCS) Score [Median (Inter-Quartile Range); unit: units on a scale] — PCS of the SF-12 is a self-reported measure of mental health-related quality of life. PCS is calculated using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
  units on a scale | 33.92 [29.05 to 44.16] | 38.32 [33.42 to 44.38] | 36.48 [31.06 to 44.37]
SF-12 Mental Component Summary (MCS) Score [Median (Inter-Quartile Range); unit: units on a scale] — MCS of the SF-12 is a self-reported measure of mental health-related quality of life. MCS is calculated using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
  units on a scale | 51.38 [45.26 to 59.24] | 50.53 [35.95 to 57.11] | 51.25 [44.94 to 57.11]

OUTCOME MEASURES:

1. Primary Outcome: Change in Epistaxis Severity Score (ESS)
Description: ESS is a standardized and reproducible outcome measure for the control of epistaxis. It is composed of six factors that are independent predictors of self-described epistaxis severity. The range is 0 to 13. The higher the score worse is epistaxis severity.
Time Frame: Baseline and month 1, month 2, month 4, month 6
Population: Participants with available data were included in the analysis.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Bevacizumab | Saline Control
Number analyzed (Participants) | 19 | 20
score on a scale
  Difference at 1 month | -2.27 [-3.27 to -1.27] | -1.16 [-2.09 to -0.24]
  Difference at 2 month | -2.27 [-3.47 to -1.07] | -1.01 [-2.13 to 0.1]
  Difference at 4 month | -2.00 [-3.30 to -0.71] | -1.16 [-2.29 to -0.02]
  Difference at 6 month | -1.34 [-2.67 to -0.01] | -0.87 [-2.05 to 0.31]
Statistical Analysis 1: Comparison: Bevacizumab vs Saline Control; Analysis between groups at month 1; Test type: Other — Linear regression model with repeated measures, controlling for patient's demographic factors, smoking status, and baseline level of ESS. The analysis is weighted by inverse probability treatment weight (IPTW); p = 0.111, Regression, Linear; Mean Difference (Net) = -1.11, 95% CI 2-sided [-2.47 to 0.26]
Statistical Analysis 2: Comparison: Bevacizumab vs Saline Control; Analysis between groups at month 2; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.131, Regression, Linear; Mean Difference (Net) = -1.26, 95% CI 2-sided [-2.9 to 0.38]
Statistical Analysis 3: Comparison: Bevacizumab vs Saline Control; Analysis between groups at month 4; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.332, Regression, Linear; Mean Difference (Net) = -0.85, 95% CI 2-sided [-2.57 to 0.88]
Statistical Analysis 4: Comparison: Bevacizumab vs Saline Control; Analysis between groups at month 6; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.597, Regression, Linear; Mean Difference (Net) = -0.48, 95% CI 2-sided [-2.25 to 1.3]

2. Secondary Outcome: Short Form-12 (SF-12) Physical Component Summary (PCS) Score
Description: PCS of the SF-12 is a self-reported measure of mental health-related quality of life. PCS is calculated using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Time Frame: Baseline and month 1, month 2, month 4, month 6
Population: Participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bevacizumab | Saline Control
Number analyzed (Participants) | 19 | 20
score on a scale
  Month 1 | 40.53 (7.78) | 40.43 (6.79)
  Month 2 | 39.71 (7.22) | 40.88 (5.3)
  Month 4 | 39.96 (7.4) | 40.71 (5.47)
  Month 6 | 39.06 (7.86) | 38.06 (6.73)
Statistical Analysis 1: Comparison: Bevacizumab vs Saline Control; Analysis between groups at month 1; Test type: Other — Linear regression model with repeated measures, controlling for patient's demographic factors, smoking status, and baseline level of PCS. The analysis is weighted by inverse probability treatment weight (IPTW); p = 0.191, Regression, Linear; Mean Difference (Net) = 2.85, 95% CI 2-sided [-1.44 to 7.13]
Statistical Analysis 2: Comparison: Bevacizumab vs Saline Control; Analysis between groups at month 2; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.914, Regression, Linear; Mean Difference (Net) = 0.29, 95% CI 2-sided [-5.02 to 5.61]
Statistical Analysis 3: Comparison: Bevacizumab vs Saline Control; Analysis between groups at month 4; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.592, Regression, Linear; Mean Difference (Net) = 1.55, 95% CI 2-sided [-4.17 to 7.28]
Statistical Analysis 4: Comparison: Bevacizumab vs Saline Control; Analysis between groups at month 6; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.31, Regression, Linear; Mean Difference (Net) = 3.1, 95% CI 2-sided [-2.92 to 9.12]

3. Secondary Outcome: Short Form-12 (SF-12) Mental Component Summary (MCS) Score
Description: MCS of the SF-12 is a self-reported measure of mental health-related quality of life. MCS is calculated using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Time Frame: Baseline and month 1, month 2, month 4, month 6
Population: Participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bevacizumab | Saline Control
Number analyzed (Participants) | 19 | 20
score on a scale
  Mean at 1 month | 51.76 (9.91) | 54.22 (6.89)
  Mean at 2 month | 54.48 (7.99) | 50.96 (8.68)
  Mean at 4 month | 51.09 (10.61) | 53.61 (7.84)
  Mean at 6 month | 48.39 (12.97) | 55.18 (8.03)
Statistical Analysis 1: Comparison: Bevacizumab vs Saline Control; Analysis between groups at month 1; Test type: Other — Linear regression model with repeated measures, controlling for patient's demographic factors, smoking status, and baseline level of MCS. The analysis is weighted by inverse probability treatment weight (IPTW); p = 0.366, Regression, Linear; Mean Difference (Net) = -2.63, 95% CI 2-sided [-8.38 to 3.11]
Statistical Analysis 2: Comparison: Bevacizumab vs Saline Control; Analysis between groups at month 2; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.816, Regression, Linear; Mean Difference (Net) = 0.82, 95% CI 2-sided [-6.12 to 7.76]
Statistical Analysis 3: Comparison: Bevacizumab vs Saline Control; Analysis between groups at month 4; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.247, Regression, Linear; Mean Difference (Net) = -4.3, 95% CI 2-sided [-11.61 to 3.02]
Statistical Analysis 4: Comparison: Bevacizumab vs Saline Control; Analysis between groups at month 6; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.035, Regression, Linear; Mean Difference (Net) = -8.18, 95% CI 2-sided [-15.76 to -0.6]

4. Secondary Outcome: Reduction in Epistaxis-related Costs (Direct and Indirect)
Description: Evaluate the effect of bevacizumab injection on direct and indirect costs in USD associated with care and management of epistaxis as well as productivity lost after treatment. The cost of caring in USD for nasal bleeding was evaluated with two surveys, the Work Productivity and Activity Impairment Questionnaire, and the HHT Costing Data Sheet.
Time Frame: Baseline, Month 2, Month 6
Population: Participants with available data are included in the analysis.
Measure: Median (Inter-Quartile Range); unit: US Dollars
Arm/Group | Bevacizumab | Saline Control
Number analyzed (Participants) | 17 | 17
US Dollars
  Baseline | 74 [41 to 678] | 16 [0 to 58]
  Month 2 | 9 [0 to 63] | 11 [0 to 617]
  Month 6 | 11 [0 to 280] | 0 [0 to 29]
Statistical Analysis 1: Comparison: Bevacizumab vs Saline Control; Analysis of intergroup difference at baseline; Test type: Other; p = 0.030, Wilcoxon rank sum test, 2-sided
Statistical Analysis 2: Comparison: Bevacizumab vs Saline Control; Analysis of intergroup difference at month 2; Test type: Other; p = 0.719, Wilcoxon rank sum test, 2-sided
Statistical Analysis 3: Comparison: Bevacizumab vs Saline Control; Analysis of intergroup difference at month 6; Test type: Other; p = 0.467, Wilcoxon rank sum test, 2-sided

ADVERSE EVENTS:
Time Frame: 6 months.
Arm/Group | Bevacizumab | Saline Control
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-08-19): https://cdn.clinicaltrials.gov/large-docs/59/NCT02389959/Prot_SAP_000.pdf